CLINICAL TRIAL: NCT06680869
Title: Early Amiodarone in Shockable Cardiac Arrest (Early-Amio) Study
Brief Title: Early Amiodarone in Shockable Cardiac Arrest
Acronym: Early-Amio
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joshua Lupton, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026455; 1K23HL173647-01 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Amiodarone Protocol (Experimental): Amiodarone administration after the second defibrillator shock, during the same two-minute cycle as the initial dose of epinephrine.
  Interventions: Drug: Amiodarone Hydrochloride Injection
- Usual Care Protocol (Active Comparator): Amiodarone administration after the third defibrillator shock, one two-minute cycle after the initial dose of epinephrine.
  Interventions: Other: Usual Care Protocol

INTERVENTIONS:
Drug: Amiodarone Hydrochloride Injection — The use of a modified treatment protocol by emergency medical services where the initial dose of amiodarone is given after the second defibrillator shock, during the same two-minute cycle as the initial dose of epinephrine, for out-of-hospital cardiac arrest due to a shockable rhythm (ventricular fibrillation or ventricular tachycardia) that is persistent or recurs after at least one defibrillation attempt.
  If an EMS agency is assigned to this arm, no downstream care after the initial dose of amiodarone is dictated by the study.
  Other Names: Early-Amiodarone Protocol
  Arms: Early Amiodarone Protocol
Other: Usual Care Protocol — The use of a usual care treatment protocol by emergency medical services where the initial dose of amiodarone is given after the third defibrillator shock, one two-minute cycle after the initial dose of epinephrine, for out-of-hospital cardiac arrest due to a shockable rhythm (ventricular fibrillation or ventricular tachycardia) that is persistent or recurs after at least one defibrillation attempt.
  If an EMS agency is assigned to this arm, no downstream care after the initial dose of amiodarone is dictated by the study.
  Arms: Usual Care Protocol

SUMMARY:
The primary objective of this pilot, pragmatic stepped-wedge cluster randomized trial is to evaluate if a modified cardiac arrest treatment algorithm calling for the administration of the initial amiodarone dose one 2-minute cycle earlier than current guidelines (during the same cycle as the initial dose of epinephrine) improves the time to amiodarone delivery in those with out-of-hospital cardiac arrest due to refractory ventricular fibrillation or ventricular tachycardia compared to usual care.

DETAILED DESCRIPTION:
The primary objective of this pilot, pragmatic stepped-wedge cluster randomized trial is to evaluate if a modified cardiac arrest treatment algorithm calling for the administration of the initial amiodarone dose one 2-minute cycle earlier than current guidelines (during the same cycle as the initial dose of epinephrine) improves the time to amiodarone delivery in those with out-of-hospital cardiac arrest due to refractory ventricular fibrillation or ventricular tachycardia compared to usual care.

The null hypothesis is that there is no difference in time to amiodarone delivery, relative to emergency medical services (EMS) arrival on-scene or time of arrest if witnessed by EMS, in the modified protocol calling for earlier amiodarone administration compared to usual care.

Evaluated secondary outcomes will include the proportion of patients receiving amiodarone before their third defibrillation, pulses present at emergency department arrival, survival to hospital discharge, neurologically intact survival at hospital discharge, timing to other critical EMS interventions, and clinical adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medical services (EMS)-treated non-traumatic out-of-hospital cardiac arrest
* Initial rhythm on EMS rhythm assessment of ventricular fibrillation or ventricular tachycardia
* Recurrence or persistence of ventricular fibrillation or ventricular tachycardia after one defibrillation attempt

Exclusion Criteria:

* Known allergy to amiodarone
* EMS-assessed contraindication to amiodarone
* Pre-existing "do-not-attempt-resuscitation" orders
* Inter-facility transportations
* Initial care by a non-participating EMS agency able to perform advanced life support interventions
* Pediatric patient as determined by EMS
* Prisoners
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 585 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Time from emergency medical services (EMS) arrival on-scene (or time of arrest if witnessed by EMS) to the administration of the initial dose of amiodarone in minutes | up to 1 day

SECONDARY OUTCOMES:
The number and proportion of patients receiving the initial dose of amiodarone from emergency medical services before the third shock from a defibrillator | up to 1 day
The number and proportion of patients with pulses present and documented by emergency medical services at the time of patient care transfer to hospital staff at emergency department arrival | up to 1 day
The number and proportion of patients surviving to be admitted to inpatient services after arrival to the emergency department | up to 1 day
The number and proportion of patients surviving to be discharged from the hospital (or 30 days, whichever is sooner) after their admission for cardiac arrest | up to 30 days
The number and proportion of patients surviving to be discharged from the hospital (or 30 days, whichever is sooner) after their admission for cardiac arrest with a Cerebral Performance Category score of 1 or 2 | up to 30 days
  The Cerebral Performance Category (CPC) score scale is 1-5:
  CPC 1: Good cerebral performance: conscious, alert, able to work, might have mild neurologic or psychologic deficit.
  CPC 2: Moderate cerebral disability: conscious, sufficient cerebral function for independent activities of daily life. Able to work in sheltered environment.
  CPC 3: Severe cerebral disability: conscious, dependent on others for daily support because of impaired brain function. Ranges from ambulatory state to severe dementia or paralysis.
  CPC 4: Coma or vegetative state: any degree of coma without the presence of all brain death criteria. Unawareness, even if appears awake (vegetative state) without interaction with environment; may have spontaneous eye opening and sleep/awake cycles. Cerebral unresponsiveness.
  CPC 5: Brain death: apnea, areflexia, EEG silence, etc.
Time from emergency medical services (EMS) arrival on-scene (or time of arrest if witnessed by EMS) to the delivery of other critical interventions in minutes | up to 1 day
  Critical interventions include: the second-fourth defibrillator shocks, the first use of double sequential external defibrillation, the administration of the first two epinephrine doses, and the time to advanced airway placement by EMS.
Number and proportion of participants with adverse events | up to 1 day
  e.g.: malignant cardiac arrhythmia, allergic reaction, recurrent cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lupton, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Sciences University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be shared with all data elements required for analysis, if de-identification is deemed feasible, with the NHLBI BioLINCC.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months from study completion. No end date.
Access Criteria: Per NHLBI BioLINCC policy

REFERENCES:
- See also: Early-Amio Study Website — https://www.ohsu.edu/school-of-medicine/emergency/early-amiodarone-shockable-cardiac-arrest-early-amio-study